CLINICAL TRIAL: NCT02912130
Title: The Multidimensional Effects of Exercise and Nutritional Interventions on Musculoskeletal Functioning, Nutritional Status and Quality of Life in Age-related Sarcopenia
Brief Title: Exercise and Nutrition Interventions in Age-related Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Hope University (Other)
Responsible Party: Principal Investigator, Omid Khaiyat, MD, PhD, Dr, Liverpool Hope University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: LiverpoolHU
Record Dates: First submitted 2016-09-12; First posted 2016-09-23 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2022-04

CONDITIONS: Sarcopenia; Muscular Atrophy
Keywords: Exercise; Nutrition; Sarcopenia; Healthy Ageing; Elderly; Muscular Hypertrophy
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): No Intervention
- Exercise (Experimental): 1. Aerobic Exercise i.e. 30-60 minutes per week of moderate intensity exercise
  2. Resistance Exercise i.e. 60 minutes per week of progressive resistance training
  Interventions: Other: Aerobic Exercise; Other: Resistance Exercise
- Exercise+Nutrition (Experimental): 1. Aerobic Exercise i.e. 30-60 minutes per week of moderate intensity exercise
  2. Dietary Supplement i.e. Protein Supplementation 1.2-1.5g/kg/body weight per day
  Interventions: Dietary Supplement: Protein Supplementation; Other: Aerobic Exercise; Other: Resistance Exercise
- Nutrition (Experimental): Dietary Supplement: Protein Supplementation i.e. 1.2-1.5g/kg/body weight per day
  Interventions: Dietary Supplement: Protein Supplementation

INTERVENTIONS:
Dietary Supplement: Protein Supplementation — 1.2-1.5g/kg/body weight per day
  Arms: Exercise+Nutrition; Nutrition
Other: Aerobic Exercise — 30-60 minutes per week of moderate intensity exercise
  Arms: Exercise; Exercise+Nutrition
Other: Resistance Exercise — 60 minutes per week of progressive resistance training
  Arms: Exercise; Exercise+Nutrition

SUMMARY:
This project will investigate the synergistic effects of Aerobic and Resistance type Exercise, in combination with Protein Supplementation, on; Body Composition, Musculoskeletal Functioning, Nutritional Status and Quality of Life in Age-related Sarcopenia.

DETAILED DESCRIPTION:
Musculoskeletal ageing is an inevitable process associated with profound morphological and functional changes that will ultimately transition an individual from independent, to dependable living, relying heavily on personal health care for survival. The United Kingdom (UK) population aged over 65 years is expected to rise from 8.8 to 11.3 million by 2025. As life expectancy increases due to advances in medical treatment, an age-related disease termed sarcopenia, has become more prevalent in the elderly. Sarcopenia, described as the loss of musculoskeletal mass, strength and/or physical functioning with age, manifests after the 6th decade and rapidly increases after the 8th decade, resulting in a deterioration of health status and quality of life. To manage the looming health and economic consequences of sarcopenia, suitable therapeutic strategies to manage the condition are warranted. Therefore, this randomised control trial (RCT) will investigate the effects of 16-weeks of exercise and nutritional interventions in inactive senior citizens (60 - 90 years old).

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants
* 60 - 90 years of age
* Resident in North West, England, UK
* BMI 18.5-30 kg/m
* Can speak and understand English
* Willing to consent and follow the study procedures

Exclusion Criteria:

* Recent (i.e. past 3 months) or concurrent participation in any clinical trial or dietary and/or exercise intervention program
* Self-reported lactose intolerance
* Uncontrolled diabetes (HbA1C >10)
* Uncontrolled Hypertension (160/100) and uncontrolled hypotension (<100 systolic)
* Treatment with Beta Blockers, Calcium Channel Blockers, Digitalis, Bronchodilator,
* Diuretics, Vasodilators
* Current hormone therapy such as insulin, testosterone or hormone replacement therapy
* History of falls/osteoporosis
* Major psychological/mental illness
* Medical conditions that precluded safe participation in an exercise program
* Other major systemic diseases: Liver and kidney diseases, Advanced gastrointestinal disorders, Cardiovascular Diseases, Advanced chronic obstructive pulmonary disease, Advanced Rheumatoid Arthritis, Cancer

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Body Composition: Lean Muscle/Fat Tissue 1) appendicular lean mass (kg) divided by height (meters-squared) and 2) appendicular lean mass divided by body mass index | 16 weeks

SECONDARY OUTCOMES:
Grip Strength: Hand Grip Dynanometer (kg) | 16 weeks
Gait speed during timed 4-meter walk (m/s) | 16 Weeks
Time to complete five chair rises (m/s) | 16 Weeks
Balance assessment: 1) feet side to side, 2) semi-tandem, 3) full tandem, and 4) single leg. Scored as Yes or No. | 16 Weeks
Isometric Strength - Knee Flexion/Extension: Dynanometer (Nm/Kg) | 16 Weeks
Muscle Fatigue: Upper & Lower limb: 25% of MVC during 60 seconds using Electromyography (EMG), measured in millivolts (mV) | 16 Weeks
Exercise Tolerance: Six Minute Walk Test (metres) | 16 Weeks
10-metre Gait analysis during habitual walking speed using Electromyography (EMG) | 16 Weeks
10-metre Gait analysis during habitual walking speed using Three-Dimensional Motion Capture - 1) Spatiotemporal, 2) Kinematics | 16 Weeks
Biochemical: Glycated Haemoglobin (HBA1c) (%) | 16 Weeks
Biochemical: C-Reactive Protein (CRP) (mg/L) | 16 Weeks
Biochemical: Insulin-Like Growth Factor 1 (IGF-1) (ng/ml) | 16 Weeks
Arterial Pressure: Pulse Wave Velocity (m/s) | 16 Weeks
Energy Balance: Periodic Food Diary (Kcal) | 16 Weeks
World Health Organization Quality Of Life Assessment (WHOQOL): Each question is scored from 1-5 on a response scale | 16 Weeks
Short-Form Health Survey (SF-12): Each question is scored between 1-6 on a response scale | 16 Weeks
Activities of Daily Living (ADL): Each response is scored as either: 0 or 1 | 16 Weeks
Mini-Mental State Examination (MMSE): Each correct response is scored as 1 point | 16 Weeks
Nutritional Status: Mini-Nutritional Assessment (MNA) - Classified as (Low, Moderate, High risk) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Omid Alizadehkhaiyat, MD, PhD, Principal Investigator — Liverpool Hope University
Locations (1):
- Liverpool Hope University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Witard OC, Wardle SL, Macnaughton LS, Hodgson AB, Tipton KD. Protein Considerations for Optimising Skeletal Muscle Mass in Healthy Young and Older Adults. Nutrients. 2016 Mar 23;8(4):181. doi: 10.3390/nu8040181. PMID 27023595
- [Background] Lourenco RA, Perez-Zepeda M, Gutierrez-Robledo L, Garcia-Garcia FJ, Rodriguez Manas L. Performance of the European Working Group on Sarcopenia in Older People algorithm in screening older adults for muscle mass assessment. Age Ageing. 2015 Mar;44(2):334-8. doi: 10.1093/ageing/afu192. Epub 2014 Dec 23. PMID 25539836
- [Background] Yu SC, Khow KS, Jadczak AD, Visvanathan R. Clinical Screening Tools for Sarcopenia and Its Management. Curr Gerontol Geriatr Res. 2016;2016:5978523. doi: 10.1155/2016/5978523. Epub 2016 Feb 4. PMID 26966433
- [Background] Churchward-Venne TA, Holwerda AM, Phillips SM, van Loon LJ. What is the Optimal Amount of Protein to Support Post-Exercise Skeletal Muscle Reconditioning in the Older Adult? Sports Med. 2016 Sep;46(9):1205-12. doi: 10.1007/s40279-016-0504-2. PMID 26894275
- [Background] Kraschnewski JL, Sciamanna CN, Poger JM, Rovniak LS, Lehman EB, Cooper AB, Ballentine NH, Ciccolo JT. Is strength training associated with mortality benefits? A 15year cohort study of US older adults. Prev Med. 2016 Jun;87:121-127. doi: 10.1016/j.ypmed.2016.02.038. Epub 2016 Feb 24. PMID 26921660
- [Background] Witard OC, McGlory C, Hamilton DL, Phillips SM. Growing older with health and vitality: a nexus of physical activity, exercise and nutrition. Biogerontology. 2016 Jun;17(3):529-46. doi: 10.1007/s10522-016-9637-9. Epub 2016 Feb 15. PMID 26878863
- [Background] Chang SF, Lin PL. Systematic Literature Review and Meta-Analysis of the Association of Sarcopenia With Mortality. Worldviews Evid Based Nurs. 2016 Apr;13(2):153-62. doi: 10.1111/wvn.12147. Epub 2016 Feb 4. PMID 26844538
- [Background] Csapo R, Alegre LM. Effects of resistance training with moderate vs heavy loads on muscle mass and strength in the elderly: A meta-analysis. Scand J Med Sci Sports. 2016 Sep;26(9):995-1006. doi: 10.1111/sms.12536. Epub 2015 Aug 24. PMID 26302881
- [Background] Xu ZR, Tan ZJ, Zhang Q, Gui QF, Yang YM. Clinical effectiveness of protein and amino acid supplementation on building muscle mass in elderly people: a meta-analysis. PLoS One. 2014 Sep 30;9(9):e109141. doi: 10.1371/journal.pone.0109141. eCollection 2014. PMID 25268791
- [Background] Komar B, Schwingshackl L, Hoffmann G. Effects of leucine-rich protein supplements on anthropometric parameter and muscle strength in the elderly: a systematic review and meta-analysis. J Nutr Health Aging. 2015 Apr;19(4):437-46. doi: 10.1007/s12603-014-0559-4. PMID 25809808
- [Background] Ko SU, Hausdorff JM, Ferrucci L. Age-associated differences in the gait pattern changes of older adults during fast-speed and fatigue conditions: results from the Baltimore longitudinal study of ageing. Age Ageing. 2010 Nov;39(6):688-94. doi: 10.1093/ageing/afq113. Epub 2010 Sep 10. PMID 20833863
- [Derived] Kirk B, Mooney K, Vogrin S, Jackson M, Duque G, Khaiyat O, Amirabdollahian F. Leucine-enriched whey protein supplementation, resistance-based exercise, and cardiometabolic health in older adults: a randomized controlled trial. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):2022-2033. doi: 10.1002/jcsm.12805. Epub 2021 Sep 14. PMID 34520104
- [Derived] Kirk B, Mooney K, Amirabdollahian F, Khaiyat O. Exercise and Dietary-Protein as a Countermeasure to Skeletal Muscle Weakness: Liverpool Hope University - Sarcopenia Aging Trial (LHU-SAT). Front Physiol. 2019 Apr 25;10:445. doi: 10.3389/fphys.2019.00445. eCollection 2019. PMID 31133863